CLINICAL TRIAL: NCT02574377
Title: Myeloid and Plasmacytoid Blood Dendritic Cells for Immunotherapy of Stage III Melanoma Patients
Brief Title: myDC/pDC in Stage III Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49528.000.14
Record Dates: First submitted 2015-09-30; First posted 2015-10-12 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

ARMS (3):
- A: myDC vaccination (Experimental): intranodal injection with tumor peptide-loaded myeloid dendritic cells
  Interventions: Drug: A: myDC vaccination
- B: pDC vaccination (Experimental): intranodal injection with tumor peptide-loaded plasmacytoid dendritic cells
  Interventions: Drug: B: pDC vaccination
- C: combined myDC/pDC vaccination (Experimental): intranodal injection with tumor peptide-loaded myeloid and plasmacytoid dendritic cells
  Interventions: Drug: C: combined myDC/pDC vaccination

INTERVENTIONS:
Drug: A: myDC vaccination
  Arms: A: myDC vaccination
Drug: B: pDC vaccination
  Arms: B: pDC vaccination
Drug: C: combined myDC/pDC vaccination
  Arms: C: combined myDC/pDC vaccination

SUMMARY:
This is an interventional study to test the immunogenicity of combined adjuvant myDC and pDC vaccination versus adjuvant myDC or pDC vaccination alone in stage III melanoma patients.

DETAILED DESCRIPTION:
Stage lll melanoma patients will receive pDC (arm A, n=10), myDC (arm B, n=10) or combined pDC/myDC (arm C, n=10). Subsequent vaccinations will be performed according to the protocol: 2 biweekly vaccinations of intranodal injections with pDC, myDC or the combination with pDC and myDC. After each vaccination the investigators will examine peripheral blood for proliferative and humoral KLH immune responses. After the vaccinations, a DTH with peptide loaded blood DC is performed from which biopsies are taken for T cell analysis. lf patients remain disease free, the investigators will repeat this cycle with a 6 months interval up to a total of three cycles. lf a tumor recurrence occurs a biopsy will be taken for laboratory evaluation.

ELIGIBILITY:
Inclusion Criteria:

* stage III melanoma
* WHO performance status 0-1
* radical lymph node dissection is schedule or performed within 12 weeks prior to start of study treatment

Exclusion Criteria:

* irresectable disease
* any concurrent adjuvant therapy
* concomitant use of oral immunosuppressive drugs
* autoimmune diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
immunogenicity - type I IFN | up to 1.5 years
  Type I IFN gene expression in PBMC shortly after vaccination. The occurrence of the type I IFN response in patients will be compared between the arms.
immunogenicity - response to KLH | up to 1.5 years
  Proliferative, effector cytokine and humoral responses to keyhole limpet hemocyanin (KLH).The occurrence of the response will be compared between the arms.
immunogenicity - T cells in DTH | up to 1.5 years
  Functional response and tetramer analysis of DTH infiltrating T cells against tumor peptides. The occurrence of the response will be compared between the arms.

SECONDARY OUTCOMES:
biodistribution/localization of pDC and myDC in the lymph node | within 1 week after vaccination 1
  biodistribution/localization of the injected labeled pDC and/or myDC in the resected lymph node by multiple techniques
safety - Toxicity will be assessed according to the NCI Common Toxicity Criteria, CTC version 4.0 | up to 1.5 years
  Toxicity will be assessed according to the NCI Common Toxicity Criteria, CTC version 4.0
quality of life | 5 years
  To assess the quality of life the EORTC QLQ-C30 questionnaire will be used.
progression-free survival | 5 years
  time from radical lymph node dissection to recurrence of (distant) disease
overall survival | 5 years
  time from radical lymph node dissection to death

CONTACTS AND LOCATIONS:
Overall Officials: Winald Gerritsen, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands